CLINICAL TRIAL: NCT00119886
Title: Botox on Vulvar Vestibulitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Bosex
Record Dates: First submitted 2005-07-06; First posted 2005-07-14 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Vulvar Vestibulitis; Vulvar Diseases
MeSH Terms: conditions — Vulvar Vestibulitis; Vulvar Diseases | interventions — Botulinum Toxins

INTERVENTIONS:
Drug: Botulinum toxin

SUMMARY:
The study seeks to evaluate the effect of botulinum toxin on vulvar vestibulitis (VVS) after local injection with Botox, a potential treatment to relieve patients of vulvar pain, reducing the need for painkillers, and improving the sexual quality of life of the patients.

DETAILED DESCRIPTION:
Vulvar vestibulitis (VVS) is characterized by pain confined to the vulvar vestibule that occurs upon touch and attempted introitus entry ( e.g. intercourse, tampon insertion), with minimal associated clinical findings.

The aetiology of VVS is not well established and many variables have been associated with the condition, e.g. neuropathy secondary to inflammation.

Injection of Botulinum Toxin is tested as a therapeutic option for this condition.

A temporary paralytic effect on the surrounding skeletal muscle hypertonicity is seen and earlier in cases described as a successful treatment of pelvic floor dysfunction, dyspareunia and interstitial cystitis.

ELIGIBILITY:
Inclusion Criteria:

* Vulvar vestibulitis
* Safe birth control

Exclusion Criteria:

* Treated earlier with Botulinum toxin
* Ongoing vulvar infection
* Age<18
* Skin disease
* Pregnancy
* Myasthenia gravis
* Amyotrophic lateral sclerosis (ALS)
* Diabetes
* Using:

  * Calcium antagonists;
  * Aminoglycosides;
  * Magnesium sulfate;
  * Systemic steroid treatment

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2005-04; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Reduce vulvar pain on a visual analogue scale (VAS).

SECONDARY OUTCOMES:
Investigate the effect on sexuality, quality of life, marital relationship, depression and need of analgesics

CONTACTS AND LOCATIONS:
Overall Officials: Christina Damsted Petersen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Result] Gunter J, Brewer A, Tawfik O. Botulinum toxin a for vulvodynia: a case report. J Pain. 2004 May;5(4):238-40. doi: 10.1016/j.jpain.2004.02.575. PMID 15162347
- See also: Related Info — http://www.nva.org/